CLINICAL TRIAL: NCT02506634
Title: The Primary Symptoms of GERD in Chinese Outpatients in Gastroenterology Department: A Cross-sectional Investigation
Brief Title: The Primary Symptoms of GERD(Gastroesophageal Reflux Disease) in Chinese Outpatients in Gastroenterology Department
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, tanniandi, Resident physician, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: ESR-14-10521
Record Dates: First submitted 2015-07-20; First posted 2015-07-23 (Estimated); Results first posted 2019-12-04 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Gastroesophageal Reflux
Keywords: symptom
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Participants with upper gastrointestinal symptoms: Participants are stratified at baseline based on their main upper gastrointestinal symptoms and then evaluated for GERD using different methods (i.e., reflux esophagitis on endoscopy or positive acid exposure time (AET) on reflux monitoring). Patients would then be given Esomeprazole MUPS（ Multiple Unit Pellet System）20 mg bid for evaluating the ability of the PPI Test for GERD. According to the guidelines, the duraion of PPI treatment was 4 weeks and 8 weeks for endoscopy negative patients and patients has reflux esophagitis, respectively.
  Interventions: Drug: Esomeprazole MUPS, 20 mg

INTERVENTIONS:
Drug: Esomeprazole MUPS, 20 mg — According to the guidelines, the PPI treatment duration would be 8 weeks(Esomeprazole MUPS, 20 mg bid) for patients with reflux esophagitis and 4 weeks (Esomeprazole MUPS, 20 mg bid) for patients with normal findings on endoscopy.
  Other Names: Nexium

SUMMARY:
Consecutive patients aged 18-65 years who go to the gastroenterology clinic presented with upper gastrointestinal discomfort would be included. All patients underwent upper endoscopy or an ambulatory 24-h pH(Potential Of Hydrogen) monitoring.Pathologic esophageal acid reflux was defined as the percentage total time for which a pH value < 4 was >4.2 % in the distal esophagus. Then, patients were treated with esomeprazole 20 mg twice daily for 28 days. The symptom scores were measured by the frequency score multiplied by the severity scores of the predominant symptom before and at the end of the treatment, and the " PPI test " was defined as positive if the overall scores of the predominant dyspeptic symptom in the fourth week decreased by >50 % compared with those of the baseline.

GERD is defined by either 24-hour impedance-pH monitoring or positive PPI(proton pump inhibitor) test or positive result from endoscopy. The percentage of each symptom of GERD in the symptom questionnaire in Chinese outpatients in Gastroenterology department will be calculated. The symptom of the highest percentage will be the primary symptom.

DETAILED DESCRIPTION:
Primary Objective：To define the primary symptom of GERD in Chinese outpatients in Gastroenterology department Secondary Objective：1. To investigate the symptom distribution of patients who present with symptoms originated from upper gastrointestinal tract and have pathologic esophageal reflux established by 24-hour impedance-pH monitoring, upper endoscopy, or proton pump inhibitor test.

2. To evaluate the life quality of patients with atypical GERD symptoms (symptoms except heartburning and regurgitation) 3. To investigate the diagnostic value of proton pump inhibitor trial to diagnose GERD with atypical reflux symptoms 4. To investigate the predictive value of Gerd Q to diagnose GERD with atypical reflux symptoms with heartburn or regurgitation

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients aged 18-65 years who go to the gastroenterology clinic presented with upper gastrointestinal discomfort, such as heartburn, regurgitation, dysphagia, substernal pain, epigastric pain, epigastric burning, early satiety, postprandial fullness.
* Whose previous symptoms should last for at least 3 months and be at least 3 days per week in frequency with moderate severity.
* Able to fill in the questionaires.

Exclusion Criteria:

* gastric or duodenal ulcers, upper GI neoplasms on upper endoscopy
* severe cardiac or pulmonary diseases, diabetes or rheumatic diseases
* history of operations in the upper GI tract
* renal failure or abnormal liver function
* use of non-steroidal anti-inflammatory drugs (NSAIDs)
* allergy to esomeprazole
* Pregnancy or lactating mother

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be done in the outpatient clinic, department of Gastroenterology, first affiliated hospital, sun yet-sen university. Consecutive patients who met the inclusion criteria in the Gastroenterology clinic in the first affiliated hospital will be enrolled in the study. There will not be any randomization in the study.
Sampling Method: Non-Probability Sample
Enrollment: 374 (Actual)
Dates: Start 2015-08; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Minhu Chen, PHD, Study Director — vice-president of the first Affiliated hospital of SYSU
Locations (1):
- the first affiliated hospital of SYSU, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zhang MY, Tan ND, Li YW, Sifrim D, Pandolfino JE, Xiao YL, Chen MH. Esophageal symptoms versus epigastric symptoms: Relevance for diagnosis of gastroesophageal reflux disease. J Dig Dis. 2020 Dec;21(12):696-704. doi: 10.1111/1751-2980.12946. Epub 2020 Nov 8. PMID 32975045

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four hundred consecutive patients with upper gastrointestinal (GI) symptoms were screened, 19 patients who didn't meet the inclusion criteria and 7 patients with major motility disorders on high resolution manometry were excluded. Thus, a total of 374 patients were finally enrolled in the current study.
Pre-assignment Details: The current study was a single Arm study where all participants with upper GI symptoms were enrolled and tested for gastro-esophageal reflux disease (GERD) via endoscopy and 24-hour reflux monitoring. Participants were then given proton pump inhibitor(PPI) treatment and the course was decided base on the endoscopy findings.
Groups:
- Patients With Upper GI Symptoms: Participants were stratified at baseline based on their main gastrointestinal symptoms and then evaluated for GERD using different methods. They also recieved PPI treatment (Esomeprazole MUPS, 20 mg, bid, 4 or 8 weeks) and finished GERDQ.
Period: Overall Study
Arm/Group | Patients With Upper GI Symptoms
Started | 374
Participants Who Were Diagnosed as GERD | 154
Participants Who Received PPI Treatment | 357
Participants Who Finished GERDQ | 342
Completed | 357
Not Completed | 17

BASELINE CHARACTERISTICS:
Population: The aim of the current study was to investigate the symptom spectrum of GERD, and patients presented with upper GI symptoms including heartburn, regurgitation, chest pain, dysphagia, epigastric pain, epigastric burning, early satiety and postprandial fullness were enrolled. Baseline analysis population was based on patients' predominant symptom.
Groups:
- Patients With Predominant Heartburn: Patients with predominant heartburn were evaluated for GERD using different methods (i.e., reflux esophagitis on endoscopy or positive acid exposure time (AET) on reflux monitoring). They also recieved PPI test and finished GERDQ.
- Patients With Predominant Regurgitation: Patients with predominant regurgitation were evaluated for GERD using different methods (i.e., reflux esophagitis on endoscopy or positive acid exposure time (AET) on reflux monitoring). They also recieved PPI test and finished GERDQ.
- Patients With Predominant Chest Pain: Patients with predominant chest pain were evaluated for GERD using different methods (i.e., reflux esophagitis on endoscopy or positive acid exposure time (AET) on reflux monitoring). They also recieved PPI test and finished GERDQ.
- Patients With Predominant Dysphagia: Patients with predominant dysphagia were evaluated for GERD using different methods (i.e., reflux esophagitis on endoscopy or positive acid exposure time (AET) on reflux monitoring). They also recieved PPI test and finished GERDQ.
- Patients With Predominant Epigastric Pain: Patients with predominant epigastric pain were evaluated for GERD using different methods (i.e., reflux esophagitis on endoscopy or positive acid exposure time (AET) on reflux monitoring). They also recieved PPI test and finished GERDQ.
- Patients With Predominant Epigastric Burning: Patients with predominant epigastric burning were evaluated for GERD using different methods (i.e., reflux esophagitis on endoscopy or positive acid exposure time (AET) on reflux monitoring). They also recieved PPI test and finished GERDQ.
- Patients With Predominant Postprandial Fullness: Patients with predominant postprandial fullness were evaluated for GERD using different methods (i.e., reflux esophagitis on endoscopy or positive acid exposure time (AET) on reflux monitoring). They also recieved PPI test and finished GERDQ.
- Patients With Predominant Early Satiety: Patients with predominant early satiety were evaluated for GERD using different methods (i.e., reflux esophagitis on endoscopy or positive acid exposure time (AET) on reflux monitoring). They also recieved PPI test and finished GERDQ.
- Total: Total of all reporting groups
Arm/Group | Patients With Predominant Heartburn | Patients With Predominant Regurgitation | Patients With Predominant Chest Pain | Patients With Predominant Dysphagia | Patients With Predominant Epigastric Pain | Patients With Predominant Epigastric Burning | Patients With Predominant Postprandial Fullness | Patients With Predominant Early Satiety | Total
Number analyzed (Participants) | 87 | 82 | 63 | 12 | 35 | 29 | 64 | 2 | 374
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.90 (12.25) | 40.96 (14.06) | 43.27 (10.70) | 41.83 (13.29) | 42.54 (14.56) | 43.83 (14.34) | 39.88 (13.31) | 30.50 (12.02) | 42.88 (12.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 40 | 32 | 7 | 24 | 18 | 31 | 2 | 196
  Male | 45 | 42 | 31 | 5 | 11 | 11 | 33 | 0 | 178
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 22.22 (3.21) | 22.07 (3.17) | 22.69 (3.42) | 21.20 (3.22) | 21.95 (3.31) | 22.78 (3.05) | 21.39 (2.81) | 17.98 (1.12) | 22.09 (3.15)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Symptom of GERD in Chinese Outpatients in Gastroenterology Department
Description: GERD can be diagnosed by more than one different criteria (i.e."reflux esophagitis on endoscopy"; "positive acid exposure time (AET) on reflux monitoring";"Either reflux esophagitis on endoscopy or positive AET on reflux monitoring") in a single participant. When different criteria was used to diagnose GERD, the percentage of GERD patients with different predominant symptom will be calculated. The symptom of the highest percentage will be the primary symptom.
Time Frame: over 3 years
Population: GERD is diagnosed based on different criteria among 374 enrolled patients, and then the percentage of GERD patients with different predominant symptom will be calculated. The symptom of the highest percentage will be the primary symptom.
Measure: Count of Participants; unit: Participants
Groups:
- GERD Patients Defined by Reflux Esophagitis on Endoscopy; GERD Patients Defined by Positive AET on Reflux Monitoring; GERD Patients Defined by Either Endoscopy or Reflux Monitoring: The percentage of GERD patients with different predominant symptom will be calculated.
Arm/Group | GERD Patients Defined by Reflux Esophagitis on Endoscopy | GERD Patients Defined by Positive AET on Reflux Monitoring | GERD Patients Defined by Either Endoscopy or Reflux Monitoring
Number analyzed (Participants) | 79 | 111 | 154
Participants
  Heartburn | 19 | 30 | 42
  Regurgitation | 23 | 30 | 38
  Chest pain | 9 | 16 | 23
  Dysphagia | 2 | 4 | 4
  Epigastric pain | 9 | 5 | 11
  Epigastric burning | 4 | 11 | 13
  Postprandial fullness | 13 | 15 | 23
  Early satiety | 0 | 0 | 0

2. Secondary Outcome: The Percentage of Participants Diagnosed With Reflux Esophagitis Using Endoscopy Among Participants With Different Main Baseline Symptoms
Description: The percentage of paticipants diagnosed with reflux esophagitis on endoscopy among patients with different main symptom in the symptom questionnaire in Chinese outpatients in Gastroenterology department will be calculated.
Time Frame: over 3 years
Population: Among 374 enrolled patients presented with different main symptom, the percentage of patients with reflux esophagitis was calculated.
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Predominant Heartburn: The percentage of paticipants diagnosed with reflux esophagitis on endoscopy among patients with predominant heartburn will be calculated.
- Patients With Predominant Regurgitation: The percentage of paticipants diagnosed with reflux esophagitis on endoscopy among patients with predominant regurgitation will be calculated.
- Patients With Predominant Chest Pain: The percentage of paticipants diagnosed with reflux esophagitis on endoscopy among patients with predominant chest pain will be calculated.
- Patients With Predominant Dysphagia: The percentage of paticipants diagnosed with reflux esophagitis on endoscopy among patients with predominant dysphagia will be calculated.
- Patients With Predominant Epigastric Pain: The percentage of paticipants diagnosed with reflux esophagitis on endoscopy among patients with predominant epigastric pain will be calculated.
- Patients With Predominant Epigastric Burning: The percentage of paticipants diagnosed with reflux esophagitis on endoscopy among patients with predominant epigastric burning will be calculated.
- Patients With Predominant Postprandial Fullness: The percentage of paticipants diagnosed with reflux esophagitis on endoscopy among patients with predominant postprandial fullness will be calculated.
- Patients With Predominant Early Satiety: The percentage of paticipants diagnosed with reflux esophagitis on endoscopy among patients with predominant early satiety will be calculated.
Arm/Group | Patients With Predominant Heartburn | Patients With Predominant Regurgitation | Patients With Predominant Chest Pain | Patients With Predominant Dysphagia | Patients With Predominant Epigastric Pain | Patients With Predominant Epigastric Burning | Patients With Predominant Postprandial Fullness | Patients With Predominant Early Satiety
Number analyzed (Participants) | 87 | 82 | 63 | 12 | 35 | 29 | 64 | 2
Participants | 19 | 23 | 9 | 2 | 9 | 4 | 13 | 0

3. Secondary Outcome: The Percentage of Participants Diagnosed With Pathological Acid Reflux Using Reflux Monitoring Among Participants With Different Main Baseline Symptoms
Description: The percentage of paticipants diagnosed with pathological acid reflux using reflux monitoring among patients with different main baseline symptom in the symptom questionnaire in Chinese outpatients in Gastroenterology department will be calculated.
Time Frame: over 3 years
Population: Among 374 enrolled patients presented with different main symptom, the percentage of patients with pathological acid reflux was calculated.
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Predominant Heartburn: The percentage of paticipants diagnosed with pathological acid reflux using reflux monitoring among patients with predominant heartburn will be calculated.
- Patients With Predominant Regurgitation: The percentage of paticipants diagnosed with pathological acid reflux using reflux monitoring among patients with predominant regurgitation will be calculated.
- Patients With Predominant Chest Pain: The percentage of paticipants diagnosed with pathological acid reflux using reflux monitoring among patients with predominant chest pain will be calculated.
- Patients With Predominant Dysphagia: The percentage of paticipants diagnosed with pathological acid reflux using reflux monitoring among patients with predominant dysphagia will be calculated.
- Patients With Predominant Epigastric Pain: The percentage of paticipants diagnosed with pathological acid reflux using reflux monitoring among patients with predominant epigastric pain will be calculated.
- Patients With Predominant Epigastric Burning: The percentage of paticipants diagnosed with pathological acid reflux using reflux monitoring among patients with predominant epigastric burning will be calculated.
- Patients With Predominant Postprandial Fullness: The percentage of paticipants diagnosed with pathological acid reflux using reflux monitoring among patients with predominant postprandial fullness will be calculated.
- Patients With Predominant Early Satiety: The percentage of paticipants diagnosed with pathological acid reflux using reflux monitoring among patients with predominant early satiety will be calculated.
Arm/Group | Patients With Predominant Heartburn | Patients With Predominant Regurgitation | Patients With Predominant Chest Pain | Patients With Predominant Dysphagia | Patients With Predominant Epigastric Pain | Patients With Predominant Epigastric Burning | Patients With Predominant Postprandial Fullness | Patients With Predominant Early Satiety
Number analyzed (Participants) | 87 | 82 | 63 | 12 | 35 | 29 | 64 | 2
Participants | 30 | 30 | 16 | 4 | 5 | 11 | 15 | 0

4. Secondary Outcome: The Life Quality of GERD Patients Who Were Diagnosed by Either Reflux Esophagitis on Endoscopy or Positive Acid Exposure Time(AET) on Reflux Monitoring and Presented With Different Main Baseline Symptoms
Description: The life quality of GERD patients with different main symptoms before PPI test will be measured via the MOS 36-item short form health survey (SF-36), in which higher scores mean a better quality of life. Its maximum score is 796.5, and the minimum score is 36.5.
Time Frame: over 3 years
Population: The analysis population for this outcome measure was patients with a GERD diagnosis by either reflux esophagitis on upper endoscopy or positive acid exposure time(AET) on reflux monitoring.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GERD Patients With Predominant Heartburn: The life quality of GERD patients with predominant heartburn will be measured via the MOS 36-item short form health survey (SF-36).
- GERD Patients With Predominant Regurgitation: The life quality of GERD patients with predominant regurgitation will be measured via the MOS 36-item short form health survey (SF-36).
- GERD Patients With Predominant Chest Pain: The life quality of GERD patients with predominant chest pain will be measured via the MOS 36-item short form health survey (SF-36).
- GERD Patients With Predominant Dysphagia: The life quality of GERD patients with predominant dysphagia will be measured via the MOS 36-item short form health survey (SF-36).
- GERD Patients With Predominant Epigastric Pain: The life quality of GERD patients with predominant epigastric pain will be measured via the MOS 36-item short form health survey (SF-36).
- GERD Patients With Predominant Epigastric Burning: The life quality of GERD patients with predominant epigastric burning will be measured via the MOS 36-item short form health survey (SF-36).
- GERD Patients With Predominant Postprandial Fullness: The life quality of GERD patients with predominant postprandial fullness will be measured via the MOS 36-item short form health survey (SF-36).
- GERD Patients With Predominant Early Satiety: The life quality of GERD patients with predominant early satiety will be measured via the MOS 36-item short form health survey (SF-36).
Arm/Group | GERD Patients With Predominant Heartburn | GERD Patients With Predominant Regurgitation | GERD Patients With Predominant Chest Pain | GERD Patients With Predominant Dysphagia | GERD Patients With Predominant Epigastric Pain | GERD Patients With Predominant Epigastric Burning | GERD Patients With Predominant Postprandial Fullness | GERD Patients With Predominant Early Satiety
Number analyzed (Participants) | 42 | 38 | 23 | 4 | 11 | 13 | 23 | 0
score on a scale | 565.04 (163.59) | 582.55 (128.87) | 606.35 (134.44) | 706.67 (18.35) | 581.15 (193.52) | 545.8 (176.79) | 618.18 (152.35) |

5. Secondary Outcome: The Sensitivity of PPI Test for Diagnosis of GERD
Description: The sensitivity of PPI test for the diagnosis of GERD in patients with typical or atypical reflux symptoms will be calculated. The presence of reflux esophagitis on upper endoscopy and/or pathological acid reflux on 24-hour pH monitoring are considered as the "gold standard" for the diagnosis of GERD.
Time Frame: over 3 years
Population: This outcome measure is the sensitivity of PPI test for GERD diagnosis, so the whole analysis population would be patients who finished PPI treatment. Note: typical reflux symptoms are heartburn and regurgitation; atypical reflux symptoms are chest pain, dysphagia, epigastric pain, epigastric burning, postprandial fullness, and early satiety.
Measure: Number; unit: Percentage of true positive
Groups:
- Patients With Typical Reflux Symptoms: The sensitivity of PPI test for the diagnosis of GERD in patients with typical reflux symptoms will be calculated.
- Patients With Atypical Symptoms: The sensitivity of PPI test for the diagnosis of GERD in patients with atypical reflux symptoms will be calculated.
Arm/Group | Patients With Typical Reflux Symptoms | Patients With Atypical Symptoms
Number analyzed (Participants) | 160 | 197
Percentage of true positive | 0.64 | 0.51

6. Secondary Outcome: The Specificity of PPI Test for Diagnosis of GERD
Description: The specificity of PPI test for the diagnosis of GERD in patients with typical or atypical reflux symptoms will be calculated. The presence of reflux esophagitis on upper endoscopy and/or pathological acid reflux on 24-hour pH monitoring are considered as the "gold standard" for the diagnosis of GERD.
Time Frame: over 3 years
Population: This outcome measure is the specificity of PPI test for GERD diagnosis, so the whole analysis population would be patients who finished PPI treatment. Note: typical reflux symptoms are heartburn and regurgitation; atypical reflux symptoms are chest pain, dysphagia, epigastric pain, epigastric burning, postprandial fullness, and early satiety.
Measure: Number; unit: Percentage of true negative
Groups:
- Patients With Typical Reflux Symptoms: The specificity of PPI test for the diagnosis of GERD in patients with typical reflux symptoms will be calculated.
- Patients With Atypical Symptoms: The specificity of PPI test for the diagnosis of GERD in patients with atypical reflux symptoms will be calculated.
Arm/Group | Patients With Typical Reflux Symptoms | Patients With Atypical Symptoms
Number analyzed (Participants) | 160 | 197
Percentage of true negative | 0.40 | 0.62

7. Secondary Outcome: The Sensitivity of GERDQ for Diagnosis of GERD
Description: The sensitivity of GERDQ for the diagnosis of GERD in patients with typical or atypical reflux symptoms will be calculated. The presence of reflux esophagitis on upper endoscopy and/or pathological acid reflux on 24-hour pH monitoring are considered as the "gold standard" for the diagnosis of GERD.
Time Frame: over 3 years
Population: This outcome measure is the sensitivity of GERDQ for GERD diagnosis, so the whole analysis population would be patients who finished GERDQ. Note: typical reflux symptoms are heartburn and regurgitation; atypical reflux symptoms are chest pain, dysphagia, epigastric pain, epigastric burning, postprandial fullness, and early satiety.
Measure: Number; unit: Percentage of true positive
Groups:
- Patients With Typical Reflux Symptoms: The sensitivity of GERDQ for the diagnosis of GERD in patients with typical reflux symptoms will be calculated.
- Patients With Atypical Symptoms: The sensitivity of GERDQ for the diagnosis of GERD in patients with atypical reflux symptoms will be calculated.
Arm/Group | Patients With Typical Reflux Symptoms | Patients With Atypical Symptoms
Number analyzed (Participants) | 153 | 189
Percentage of true positive | 0.84 | 0.43

8. Secondary Outcome: The Specificity of GERDQ for Diagnosis of GERD
Description: The specificity of GERDQ for the diagnosis of GERD in patients with typical or atypical reflux symptoms will be calculated. The presence of reflux esophagitis on upper endoscopy and/or pathological acid reflux on 24-hour pH monitoring are considered as the "gold standard" for the diagnosis of GERD.
Time Frame: over 3 years
Population: This outcome measure is the specificity of GERDQ for GERD diagnosis, so the whole analysis population would be patients who finished GERDQ. Note: typical reflux symptoms are heartburn and regurgitation; atypical reflux symptoms are chest pain, dysphagia, epigastric pain, epigastric burning, postprandial fullness, and early satiety.
Measure: Number; unit: Percentage of true negative
Groups:
- Patients With Typical Reflux Symptoms: The specificity of GERDQ for the diagnosis of GERD in patients with typical reflux symptoms will be calculated.
- Patients With Atypical Symptoms: The specificity of GERDQ for the diagnosis of GERD in patients with atypical reflux symptoms will be calculated.
Arm/Group | Patients With Typical Reflux Symptoms | Patients With Atypical Symptoms
Number analyzed (Participants) | 153 | 189
Percentage of true negative | 0.24 | 0.63

ADVERSE EVENTS:
Time Frame: over 3 years
Groups:
- Patients Who Received PPI Treatment: The frequency of adverse events among patients who received PPI treatment was calculated.
Arm/Group | Patients Who Received PPI Treatment
All-Cause Mortality (participants affected / at risk) | 0/357
Serious Adverse Events (participants affected / at risk) | 1/357
Other Adverse Events (participants affected / at risk) | 42/357
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Who Received PPI Treatment (N=357)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) — There was one serious adverse event (SAE) that a patient had pneumothorax during the treatment phase and withdrew from the study, which had no causality with any drug or study procedure.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Who Received PPI Treatment (N=357)
Abdominal pain (Gastrointestinal disorders) | 11
Abdominal distension (Gastrointestinal disorders) | 10
Diarrhea (Gastrointestinal disorders) | 9
Bitter taste (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 6
Nausea (Gastrointestinal disorders) | 5
Headache (General disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-08): https://cdn.clinicaltrials.gov/large-docs/34/NCT02506634/Prot_SAP_000.pdf